CLINICAL TRIAL: NCT00541437
Title: An Open-Label Study to Investigate the Efficacy and Safety of Type 2 Diabetes Patients Switched From Sulfonylurea With Metformin to Glyburide/Metformin Combination Tablet
Brief Title: Type 2 Diabetes Patients Switched From Sulfonylurea With Metformin to Glyburide/Metformin Combination Tablet
Status: Completed | Type: Observational
Sponsor: Genovate Biotechnology Co., Ltd., (Industry)
Other Study IDs: GBL L-13
Record Dates: First submitted 2007-10-08; First posted 2007-10-10 (Estimated); Last update posted 2007-10-10 (Estimated); Status verified 2007-10

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Change from baseline of HbA1c after 16 weeks of treatment; Change from baseline of FPG after 16 weeks of treatment; Change from baseline of diabetes self-care scale by patient on drug administration after 16 weeks of treatment
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To evaluate the efficacy and safety of type 2 diabetes patients switched from sulfonylurea co-administered with metformin to glyburide/metformin combination tablet. It is expected that safety and efficacy of GlucoMet® is not inferior to co-administration of sulfonylurea and metformin.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age between 20 to 75 years and were diagnosed with type-2 DM for a minimum of 4 months before baseline.
* Maintain stable dose of sulfonylurea and metformin co-administered 4 months before baseline.
* Consider suitable to switch from current therapeutic dose to one of the eight testing regimens.
* FPG of 80-200mg/dl at screening visit
* 6.5% ≦ HbA1c ≦ 9% at screening visit, and change of HbA1c ≦ 1% within 12 weeks before screening visit.
* The body index must be between 18.5 and 35 Kg/m2 at screening visit.
* Sign and date the Informed Consent Form

Exclusion Criteria:

* Renal disease or renal dysfunction (e.g. serum creatinine > 1.5mg/dl)
* Currently significant GI disorder (such as peptic ulcer or diarrhea requiring chronic medical treatment) or which may interfere with absorption of the study drugs.
* History or concurrent liver disease or hepatic impairment (total bilirubin above upper normal limit, ALT or AST above 2.5 times of upper normal limit at screening visit.)
* Acute or chronic metabolic acidosis, including lactic acidosis, diabetic ketoacidosis, with or without coma.
* History of cardiovascular collapse (shock) or congestive heart failure (function class III to IV).
* History of stroke, myocardial infarction, coronary revascularization, or arrhythmia that requires medical treatment, within past 6 months.
* Having proliferative retinopathy.
* Current acute infection, including systemic infection with fever and/or sepsis, or pulmonary infection, cellulitis, etc.
* Having been treated with insulin during past 6 months, or treated with acarbose or glitazones with change of daily dose past 4 months.
* Seriously dehydrated.
* History of alcoholism (all the time or short-term heavy drinking) or drug abuse, or taking other investigational drug.
* Pregnant or breast feeding women or planning a pregnancy.
* Having a surgery within 4 weeks prior to entering the study or a history of cancer within five years.
* Known hypersensitive to glyburide or metformin hydrochloride.
* Any clinical condition or significant concurrent disease judged by the investigator to complicate the evaluation of the study treatment.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2006-05; Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tien-Shang Huang, M.D, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan university hospital, Taipei, Taiwan